CLINICAL TRIAL: NCT04403165
Title: Locus-coeruleus Function in Normal Elderly and AD Risk
Acronym: LEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-00002; 1R21AG067549-01 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitively Normal (CN) Older Adults (Experimental)
  Interventions: Procedure: Nocturnal polysomnography (NPSG); Procedure: Lumbar Puncture (LP); Other: PET-MR measurement with a norepinephrine transporter (NET)-selective radiotracer (S,S)-[11C]Omethylreboxetine ([11C]MRB); Behavioral: Psychomotor Vigilance Task (PVT)

INTERVENTIONS:
Procedure: Nocturnal polysomnography (NPSG) — Nocturnal polysomnography (NPSG) to measure REM sleep and sleep spindles characteristics.
Procedure: Lumbar Puncture (LP) — Lumbar puncture (LP) to measure CSF P-Tau, T-Tau and Aβ42/40 ratio.
Other: PET-MR measurement with a norepinephrine transporter (NET)-selective radiotracer (S,S)-[11C]Omethylreboxetine ([11C]MRB) — PET-MR measurement with a norepinephrine transporter (NET)-selective radiotracer (S,S)-[11C]O-methylreboxetine ([11C]MRB) to measure NET availability.
Behavioral: Psychomotor Vigilance Task (PVT) — Psychomotor vigilance task (PVT) and the OddBall to measure test taskattention performance.

SUMMARY:
Growing evidence suggests that Alzheimer's disease (AD) pathological changes begin decades before clinical symptoms and tau abnormalities in the locus coeruleus (LC) can be observed since midlife. We have previously demonstrated functional vulnerability of the LC to aging and stress, as well as an association between higher cerebrospinal fluid (CSF) tau and impaired sleep phenomena influenced by the LC. We now aim to test whether LC dysfunction can be measured in preclinical AD stages by LC targeted imaging, and whether it objectively affects sleep architecture and attention. We will test this hypothesis in 30 cognitively normal older adults by performing a full clinical evaluation, one night of polysomnography, a lumbar puncture to obtain cerebrospinal fluid, [11C]MRB PET-MR, and attention testing. This study has the potential to identify a new mechanism by which tau pathology contributes to sleep and attention dysfunction and may provide a new therapeutic target for AD prevention.

DETAILED DESCRIPTION:
The purpose of this study is three-fold: to test whether lower NET availability in the LC is associated with: first, CSF tau levels typical of preclinical stages of AD (Aim 1); second, reduced REM and spindle density (Aim 2); and third, impaired performance on attention tasks (Aim 3). The goal is to test the overarching hypothesis that LC dysfunction occurs in preclinical AD stages, can be measured with MRB-PET, and translates into impairment of sleep architecture (LC tonic dysfunction) and attention (LC phasic dysfunction).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with normal cognition and 55-75 years of age will be enrolled.
* Subjects will be within normal limits on neurological and psychiatric examinations.
* All subjects enrolled will have a CDR of 0. This will be evaluated through a clinical interview administered by a study physician (informant interview will not be required).
* All subjects will have had a minimum of 12 years of education.

Exclusion Criteria:

* History of brain tumor, MRI evidence of brain damage or brain disease including significant trauma, hydrocephalus, seizures, stroke, mental retardation or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders).
* Significant history of alcoholism or drug abuse.
* Significant history of psychiatric illness (e.g., schizophrenia, bipolar, PTSD, or life-long history of major depression).
* Geriatric Depression Scale (short form)>6.
* Insulin dependent diabetes.
* Evidence of clinically relevant cardiac, pulmonary, endocrine or hematological conditions.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging.
* History of a first-degree family member with early onset (age <60 years) dementia.
* Irregular sleep-wake rhythms (based on the actigraphy recordings) or significant OSA (AHI4%≥15).
* Taking Coumadin/warfarin and/or medications affecting cognition or sleep.
* Failure to complete all study visit within 4 months

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Methylreboxetine (MRB)-LC Mean Standardized Uptake Value Ratio (SUVR) Values | Visit 4 (1-4 weeks after LP)
Total Rapid Eye Movement (REM) Duration (Min) | Visit 3 (1-4 weeks after Visit 2)
  REM sleep is derived from in-laboratory nocturnal polysomnography (NPSG) sleep study.
Percentage of Time Spent in REM Sleep | Visit 3 (1-4 weeks after Visit 2)
  REM sleep is derived from in-laboratory nocturnal polysomnography (NPSG) sleep study.
REM Sleep Continuity | Visit 3 (1-4 weeks after Visit 2)
  Reported as percentage of REM runs that are less than 5, greater than or equal to 5 and greater than or equal to 10 minutes.
Number of sleep spindles that occur per minute during the N2 stage of sleep (N2 Spindle Density) | Visit 3 (1-4 weeks after Visit 2)
  N2 Spindle Density is derived from in-laboratory nocturnal polysomnography (NPSG) sleep study.
Mean Psychomotor Vigilance Test (PVT) Reaction Time | Visit 3 (1-4 weeks after Visit 2)
  PVT measures the reaction speed to a randomly time-occuring visual stimuli, allowing the assessment of several aspects of attention including response times, attention lapses and false starts.
Mean picture test response time | Visit 3 (1-4 weeks after Visit 2)
  The "Picture" test is used to measure the strength of the participants' memory by using a series of images. Before sleep, participants identify whether or not the image was inside or outside and whether or not the picture was emotional or neutral to them. After sleep, the participant will be shown images where some are new and some are old and asked whether or not they saw them before sleep. The images are selected from The International Affective Picture System.
Percentage of Correct Responses on the picture test | Visit 3 (1-4 weeks after Visit 2)
  The "Picture" test is used to measure the strength of the participants' memory by using a series of images. Before sleep, participants identify whether or not the image was inside or outside and whether or not the picture was emotional or neutral to them. After sleep, the participant will be shown images where some are new and some are old and asked whether or not they saw them before sleep. The images are selected from The International Affective Picture System.

SECONDARY OUTCOMES:
Levels of Hyperphosphorylated Tau (P-Tau, T-Tau) | Visit 4 (1-4 weeks after LP)
  Levels will be derived from the CSF and reported in pg/mL

OTHER OUTCOMES:
Aβ42/Aβ40 Ratio | Visit 4 (1-4 weeks after LP)
  The presence of amyloid plaques will be represented as the binary indicator of a CSF Aβ42/Aβ40 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Osorio, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Grossman School of Medicine, New York, New York
  - Icahn School of Medicine Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: The investigator who proposed to use the ricardo.osorio@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT04403165/ICF_000.pdf